CLINICAL TRIAL: NCT04386980
Title: A Phase 3, Randomized, Multi-center, Blinded, Placebo-controlled Study to Evaluate the Efficacy and Safety of Intra-articular Resiniferatoxin Versus Placebo to Manage Pain in Patients With Osteoarthritis of the Knee Whose Total Knee Replacement Surgery is Delayed
Brief Title: Study to Evaluate Resiniferatoxin in Patients With Knee Osteoarthritis Whose Total Knee Replacement Surgery is Delayed
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: To be replaced by a different protocol
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STI-RTX-3004
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Osteoarthritis, Knee; Osteo Arthritis Knee; Knee Pain Chronic
Keywords: osteoarthritis; knee pain
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — resiniferatoxin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Resiniferatoxin (Experimental): 12.5 ug of Resiniferatoxin in 5 mL volume administered once intra-articularly
  Interventions: Drug: Resiniferatoxin
- Placebo (Placebo Comparator): 5 mL of diluent in normal saline administered once intra-articularly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Resiniferatoxin — Resiniferatoxin is a compound purified from natural sources.
  Other Names: RTX
  Arms: Resiniferatoxin
Drug: Placebo — Diluent in normal saline
  Arms: Placebo

SUMMARY:
Efficacy and safety study of resiniferatoxin versus placebo to manage pain in patients with knee osteoarthritis whose TKR surgery is delayed

DETAILED DESCRIPTION:
This study evaluates the efficacy and safety of intra-articular resiniferatoxin (RTX) versus placebo to manage pain in patients with osteoarthritis of the knee whose Total Knee Replacement surgery is delayed.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent and comply with the study
* Diagnosis of osteoarthritis (OA) in the index knee
* Combined WOMAC A (pain) and C (function) subscale score of ≥ 23 at screening, using the WOMAC 5-point Likert scale
* Eligible for total knee replacement (TKR) surgery but unable to schedule surgery or undergo scheduled surgery
* In good general health; American Society of Anesthesiologists (ASA) physical status category ≤3
* Willing to use contraception for at least 30 days after receiving the study drug
* Able to understand and complete study-related forms and adequately communicate with the Investigator and site staff

Exclusion Criteria:

* Pre-existing osteonecrosis, subchondral insufficiency fracture, or knee pain attributable to disease other than OA which may confound the ability to assess response to treatment
* Concurrent medical or arthritic conditions that could interfere with evaluation of the index knee joint including, metabolic diseases, gout/pseudogout, hemochromatosis, acromegaly, fibromyalgia, rheumatoid arthritis, or other inflammatory arthropathies affecting the knee joint
* Participants with significant pain in the back or other joints (ex. hip pain) which may confound discrimination of pain assessment in index knee, as judged by the Investigator
* Undergone arthroscopic surgery of the index knee within 6 months of study drug administration, or open surgery to the index knee within 24 months of study drug administration
* Undergone replacement surgery of the index knee
* Presence of surgical hardware or other foreign bodies in the index knee
* Index knee injections with corticosteroids within 30 days, or hyaluronic acid within 3 months, or platelet-rich plasma within 6 months prior to study drug administration.
* Concurrent use of opioids for indications other than knee pain
* Arterial or venous thrombi (including stroke), myocardial infarction, hospital admission for unstable angina, cardiac angioplasty, or stenting within 12 months prior to Screening.
* Sensory peripheral neuropathy in the distal aspect of the target limb that is of moderate severity or higher at Screening
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome-related illness, acute or history of chronic hepatitis B or hepatitis C; positive tests for HIV-1 or -2 antibodies, hepatitis B surface antigen, or hepatitis C antibodies
* Specified laboratory abnormalities within 1 week of study drug administration
* History within the past 2 years of substance abuse, including alcohol
* Allergy or hypersensitivity to chili peppers, capsaicin, resiniferatoxin, acetaminophen, tramadol, radiographic contrast agents, or any of the agents to be used for sedation, anesthesia or nerve block on the day of study drug administration
* Female participants who are pregnant, planning on becoming pregnant within 30 days of receiving study drug, or are breastfeeding at Screening
* Any medical condition or medical comorbidities that, in the Investigator's opinion, could adversely impact study participation or safety, conduct of the study, or interfere with pain assessments
* Participated in a clinical study of an investigational drug within 4 half-lives of Screening or are scheduled to receive an investigational agent (therapy or device) while participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in WOMAC pain and function subscales combined score | Baseline to Week 12
  Change in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) 3.1 numerical rating scale (NRS) [0-10 scale] Pain and Function combined score. The combined score ranges from 0 to 220; a higher score indicates greater severity of disease.

SECONDARY OUTCOMES:
Safety of RTX: Incidence and severity of adverse events | Baseline through Week 12
  Incidence and severity of adverse events
Change in analgesic usage | Baseline to Week 4, Week 8, Week 12
  Change in analgesic medication usage as reported by subjects
Change in WOMAC pain and function subscales combined score | Baseline to Week 4, Week 8
  Change in the WOMAC 3.1 NRS [0-10 scale] Pain and Function combined score. The combined score ranges from 0 to 220; a higher score indicates greater severity of disease.
Patient Global Impression of Change (PGIC) in index knee pain | Baseline to Week 4, Week 8, Week 12
  Rating of change in index knee pain using the 7-point PGIC scale where 1 = very much improved and 7 = very much worsened.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Luchi, MD, Study Director — Sorrento Therapeutics, Inc.

IPD SHARING:
Plan to Share IPD: No